CLINICAL TRIAL: NCT07056959
Title: Efficacy of Collagen Matrix for Peri-implant Soft Tissue Phenotype Modification: A Randomized Controlled Trial
Brief Title: Efficacy of Collagen Matrix for Peri-implant Soft Tissue Phenotype Modification
Acronym: XCM versus FGG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed Bin Rashid University of Medicine and Health Sciences (Other)
Responsible Party: Principal Investigator, Maanas Shah, Assistant Professor, Mohammed Bin Rashid University of Medicine and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBRU-HBMCDM-RG2025-02; MBRU-HBMCDM-RG2025-02 (Other Grant/Funding Number: 2025 HBMCDM Internal Research Grant)
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-06

CONDITIONS: Keratinized Mucosa; Keratinized Tissue
Keywords: keratinized mucosa; implants; soft tissue augmentation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group - Mucograft (Experimental): XCM (Mucograft©, Geistlich Pharma® AG, Wolhusen, Switzerland) when placed at the time of healing abutment connection and its impact on peri-implant soft tissue phenotype modification
  Interventions: Procedure: Soft tissue substitute for peri-implant phenotype modification
- Control Group - Free gingival graft (Active Comparator): Use of Free gingival graft placed at the time of healing abutment connection and its impact on peri-implant soft tissue phenotype modification
  Interventions: Procedure: Control Group - Free gingival graft for soft tissue augmentation

INTERVENTIONS:
Procedure: Soft tissue substitute for peri-implant phenotype modification — XCM (Mucograft©, Geistlich Pharma® AG, Wolhusen, Switzerland) placed at the time of healing abutment connection and its impact on peri-implant soft tissue phenotype modification when
  Arms: Test group - Mucograft
Procedure: Control Group - Free gingival graft for soft tissue augmentation — Free gingival graft around implants placed at the time of healing abutment connection and its impact on peri-implant soft tissue phenotype modification
  Arms: Control Group - Free gingival graft

SUMMARY:
A stable band of keratinized mucosa (KM) around dental implants is thought to minimize tissue recession and provide resistance against mechanical, chemical, and microbial challenges, thereby preserving peri-implant tissue health. Soft tissue augmentation is often employed to enhance the soft tissue phenotype in such cases. While autogenous grafts such as free gingival grafts (FGG) remain the gold standard, xenogeneic collagen matrices (XCM) have emerged as promising alternatives, offering reduced patient morbidity and surgical time. This randomized controlled clinical trial aims to compare the clinical efficacy and patient-reported outcome measures (PROMs) of XCM versus FGG for soft tissue phenotype modification when performed during healing abutment connection around dental implants, with evaluations at both short-term (6 months) and long-term (1 and 2 years) intervals.

Thirty participants will be recruited at Dubai Health Dental Hospital and randomly assigned to receive either XCM (test) or FGG (control) augmentation. Clinical assessments will be conducted at baseline (T0), 2 weeks (T2w), and at 1 (T1), 3 (T3), 6 (T6), 12 (T12), and 24 (T24) months post-surgery.

The primary outcome is the change in KM width, measured from the mucosal margin to the mucogingival junction. Secondary outcomes include KM thickness, supracrestal tissue height, and soft tissue dimensional changes, assessed using intraoral scans (Trios 5) and superimposed STL files. Additional measurements include peri-implant soft tissue level and phenotype.

PROMs will be recorded in the first postoperative week and at the 3-year mark using a visual analog scale (VAS). Clinical indices such as plaque index, bleeding index, and probing depth will be evaluated at 6 months, 1 year, and 2 years. Marginal bone level changes and implant survival rates will also be tracked throughout the study period.

DETAILED DESCRIPTION:
A stable band of keratinized mucosa (KM) around dental implants is believed to aid in minimizing tissue recession and provide resistance to mechanical, chemical, and biological challenges, thereby supporting the health of the surrounding hard and soft tissues. The evidence regarding the effect of KM on peri-implant health in animals is conflicting. Warrer et al. concluded that the presence of KM significantly reduced mucosal recession (MR) and attachment loss (AL), while Strub et al. observed no differences in recession or bone loss of peri-implant tissues between implants with and without adequate KM. Human studies evaluating the effect of KM on various peri-implant health-related parameters, have concluded that a lack of adequate KM around dental implants is associated with more plaque accumulation, tissue inflammation, MR, and AL. Moreover, since A stable band of keratinized mucosa (KM) around dental implants is believed to aid in minimizing tissue recession and provide resistance to mechanical, chemical, and biological challenges, thereby supporting the health of the surrounding hard and soft tissues. The evidence regarding the effect of KM on peri-implant health in animals is conflicting. Warrer et al. concluded that the presence of KM significantly reduced mucosal recession (MR) and attachment loss (AL), while Strub et al. (1991) observed no differences in recession or bone loss of peri-implant tissues between implants with and without adequate KM . Human studies evaluating the effect of KM on various peri-implant health-related parameters, have concluded that a lack of adequate KM around dental implants is associated with more plaque accumulation, tissue inflammation, MR, and AL. Moreover, since most patients do not consistently adhere to supportive peri-implant maintenance programs, it is important to evaluate the role of peri-implant soft tissue characteristics in the development of peri-implant diseases. A cross-sectional study examining the significance of KM on peri-implant and adjacent natural teeth was conducted on erratic peri-implant maintenance compliers. Implant sites with KM band width of <2mm have been associated with significantly poorer clinical and radiographic parameters, suggesting a higher risk for peri-implant diseases. In response to this, a consensus report from the DGI/SEPA/Osteology Workshop emphasized the importance of measuring KM width as a part of the routine oral examination of peri-implant hard and soft tissues. In addition, if the prosthesis obstructs the identification of the peri-implant mucosal margin, its removal may be considered. Moreover, Implants with insufficient KM width require enhanced maintenance care, as they are more susceptible to plaque buildup and the development of peri-implant mucosal inflammation.

Soft tissue augmentation procedures are often implemented to improve the peri-implant soft tissue phenotype, namely the KM width, KM thickness, and supracrestal tissue height. Similar to natural teeth, soft tissue augmentation methods around implants have included autogenous techniques such as bilaminar- or apically positioned flap (APF) either alone or in combination with free gingival grafts (FGG), and connective tissue grafts (CTG). These approaches have demonstrated favourable medium to long term outcomes. Although autogenous grafts are still considered the gold standard for soft tissue augmentation procedures, a secondary interventional site for graft harvesting increases patients' morbidity. Additional intra and postoperative complications such as palatal bleeding, edema, infection, and sometimes necrosis has also been identified. Moreover, postoperative pain perception following palatal graft harvesting worsened and required additional treatment of the wound site to minimize discomfort and the need for analgesics. Additionally, the effectiveness of soft tissue augmentation may be limited by the availability of connective tissue at the donor site, particularly in cases requiring augmentation for deep horizontal alveolar defects or extensive edentulous gaps. To overcome these shortcomings, acellular dermal matrix (ADM) or xenogeneic collagen matrix (XCM) have been developed that may be associated with reduced pain perception, reduced surgery time, as they do not require an additional surgical site. While short term primary outcomes of achieving adequate zone of KM using these soft tissue substitutes have been comparable to those achieved with autogenous grafts, the efficacy of soft tissue augmentation procedures aimed at modifying the peri-implant soft tissue phenotype and their impact on peri-implant health have remained inconclusive . The network meta-analysis of randomized controlled trials demonstrated that bilaminar approaches involving CTG or ADM obtained the highest amount of KM gain, whereas APF in combination with FGG was the most effective technique for increasing KM width. KM augmentation via APF alone was associated with a significant reduction in peri-implant parameters like probing depths and plaque index, regardless of the soft tissue grafting material used, whereas bilaminar techniques with CTG or XCM showed beneficial effects on marginal bone level stability. The non-inferiority of XCM as compared to CTG or ADM have also been evaluated in various multi-center randomized controlled trials. Soft tissue augmentation with a cross-linked porcine-derived XCM at the time of implant placement showed substantial shrinkage of about 75% in areas between augmentation and 1-year follow-up. Overall, while 25% of the original soft tissue defect was eliminated by augmentation, XCM was deemed safe with no postoperative complications and limited marginal bone loss . Also, there is no consensus comparing the effectiveness of autogenous grafts and soft-tissue substitutes in achieving a stable, non-mobile peri-implant mucosa, which should be a key objective of these surgical procedures . Furthermore, there is no evidence regarding patient's preferences, studies assessing aesthetic outcomes have shown that soft tissue substitutes tend to deliver better results than FGG. However, no significant differences were observed when compared to CTG.

The timing of soft tissue augmentation around implants is a crucial factor, that may influence the choice of graft material, based on type of defect, quality and quantity of residual soft tissue and clinician's preference. The procedure is commonly performed before or at the time of implant placement, at the time of healing abutment connection or after final restorative phase. Soft tissue augmentation prior to implant placement or at healing abutment connection are considered the gold standard time points, due to the possibility of achieving complete coverage of the graft material through adequate tissue handling. Conversely, augmentation procedures at the time of implant placement or after crown delivery appears to be less predictable due to the different healing approaches and the unexpected shrinkage that may occur.

While the effectiveness of the XCM (Mucograft©, Geistlich Pharma® AG, Wolhusen, Switzerland) as a substitute for FGG around implants has been confirmed, its impact on peri-implant soft tissue phenotype modification when placed at the time of healing abutment connection requires further validation.

The aim of this randomized clinical trial is to evaluate clinical efficacy and patient-reported outcome measures (PROMs) of XCM compared to FGG for phenotype modification when conducted at time of healing abutment connection around dental implants over a short -term (6 months) and a long term (1- and 2- years) follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 or over.
* Insufficient KM width (< 2 mm) at the buccal aspect of implants at time of healing abutment placement, either for single anterior or posterior implants.
* Controlled oral hygiene (full-mouth plaque and bleeding scores ≤ 25% at baseline).
* Good compliance and commitment to attend follow-up review appointments.
* Willing to provide informed consent.

Exclusion Criteria:

* Smoking
* Untreated localized or generalized periodontal diseases
* Uncontrolled systemic diseases
* Long term use of non-steroidal anti-inflammatory medications
* History of malignancy, radiotherapy or chemotherapy
* Collagen allergy
* History of mucogingival surgery

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Changes in Keratinized Mucosa width | 6 months
  Changes in KM width - as measured from the free mucosal margin to the mucogingival junction at the mid-buccal aspect of the implant abutment or crown with a UNC-15 probe; at the follow-up time point relative to the baseline at T0

SECONDARY OUTCOMES:
Changes in KM thickness and supracrestal tissue height | 6 months
  calculating percentage of KM width (shrinkage), KM thickness and supracrestal tissue attachment reduction at the follow-up time point relative to the baseline at T0.

OTHER OUTCOMES:
Patient reported outcome measures (PROMs) | 6 months
  PROMs will be assessed during the first week post-surgery and at the 3-year follow-up using a visual analog scale (VAS) with scores ranging from 0 to 100. First week post-surgery, patients will be asked to complete a questionnaire on days 1 and 7 to evaluate post-surgical morbidity, including pain, swelling, and bleeding as well as to record the dosage of analgesics. At the 6 months follow-up, the patients will be asked to assess their comfort, satisfaction with the color and shape of the grafted area, willingness for retreatment, and overall satisfaction, all using the VAS.

CONTACTS AND LOCATIONS:
Locations (1):
- Dubai Dental Hospital, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will be made available upon reasonable request at the time of publication, in accordance with ICMJE guidelines

REFERENCES:
- [Result] Sanz M, Lorenzo R, Aranda JJ, Martin C, Orsini M. Clinical evaluation of a new collagen matrix (Mucograft prototype) to enhance the width of keratinized tissue in patients with fixed prosthetic restorations: a randomized prospective clinical trial. J Clin Periodontol. 2009 Oct;36(10):868-76. doi: 10.1111/j.1600-051X.2009.01460.x. Epub 2009 Aug 12. PMID 19678861
- [Result] Naenni N, Bienz SP, Benic GI, Jung RE, Hammerle CHF, Thoma DS. Volumetric and linear changes at dental implants following grafting with volume-stable three-dimensional collagen matrices or autogenous connective tissue grafts: 6-month data. Clin Oral Investig. 2018 Apr;22(3):1185-1195. doi: 10.1007/s00784-017-2210-3. Epub 2017 Sep 18. PMID 28924826
- [Result] Cosyn J, Eeckhout C, De Bruyckere T, Eghbali A, Vervaeke S, Younes F, Christiaens V. A multi-centre randomized controlled trial comparing connective tissue graft with collagen matrix to increase soft tissue thickness at the buccal aspect of single implants: 1-year results. J Clin Periodontol. 2022 Sep;49(9):911-921. doi: 10.1111/jcpe.13691. Epub 2022 Jul 20. PMID 35781692